CLINICAL TRIAL: NCT05986097
Title: The Breakfast Study: A Small Steps, Low-literacy, Breakfast-focused Dietary Self-management Intervention for Adults With Poorly Controlled Type 2 Diabetes
Brief Title: The Breakfast Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Laura Saslow, Associate Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00225646
Record Dates: First submitted 2023-07-17; First posted 2023-08-14 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes
Keywords: Very low carbohydrate diet; Nutrition therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Breakfast

STUDY DESIGN:
Intervention Model Description: All participants will be provided the same intervention.
Masking Description: Blood tests and continuous glucose monitoring are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Very low-carbohydrate breakfast (Experimental): Materials will encourage eating a very low-carbohydrate breakfast (or first meal of the day), with no more than about 5-10 non-fiber (net) grams of carbohydrates each.
  Interventions: Behavioral: Breakfast

INTERVENTIONS:
Behavioral: Breakfast — We will provide participants recipes and information to support this dietary change.

SUMMARY:
The investigators will conduct an acceptability, feasibility, preliminary effectiveness trial of a 4-month, online, very low-carbohydrate breakfast-focused program in 120 adults with type 2 diabetes. The investigators will measure acceptability and feasibility, plus critical efficacy outcomes, such as changes in HbA1c, anti-hyperglycemic medications, glycemic variability, body weight, blood pressure, and lipids.

DETAILED DESCRIPTION:
More than 15% of U.S. adults with type 2 diabetes have poorly controlled blood gluocse, here defined as a glycated hemoglobin (HbA1c) level of 7.0% or higher. These adults have an elevated health risk of a variety of outcomes, including amputation and mortality from cardiovascular disease and from all causes. Nutrition- focused interventions can be effective for improving glycemic control, reducing anti-hyperglycemic medications, and reducing body weight, all of which are critical outcomes for adults with type 2 diabetes. However, typical nutrition-focused interventions can be burdensome, often requiring complex instructions and a complete overhaul of one's diet. Additionally, adults with poorly controlled type 2 diabetes are more likely to have low literacy levels, which can be a barrier for adherence to complex interventions. Therefore, an effective intervention for adults with poorly controlled diabetes who may have lower health literacy levels is necessary to reduce both HbA1c levels and anti-hyperglycemic medications. Carbohydrate intake has the strongest impact on post-prandial glycemia of any dietary factor, and a very low-carbohydrate diet-due to its ability to improve glycemic control-is now recommended by the American Diabetes Association (ADA) for the treatment of type 2 diabetes. The investigators hypothesize that some of the benefits of a very low-carbohydrate diet may be available to individuals who change only their breakfasts to be very low-carbohydrate, rather than modifying their entire diet.

Thus, the investigators will conduct an acceptability, feasibility, preliminary effectiveness trial of a 4-month, online, small- steps, low-literacy, very low-carbohydrate breakfast-focused program in 120 adults with poorly controlled type 2 diabetes. The investigators will measure acceptability and feasibility, plus critical efficacy outcomes, such as changes in HbA1c, anti-hyperglycemic medications, glycemic variability, body weight, blood pressure, and lipids.

The investigators will also test whether factors such as sex, health literacy level, and baseline insulin resistance significantly moderate the impact of the intervention on change in HbA1c and change in anti-hyperglycemic medications.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c 7% or higher
* 18-80 years old
* The ability to understand verbal and written English
* Willingness to follow the prescribed diet
* Able to consent and follow directions
* Willingness to regularly check blood glucose levels as required

Exclusion Criteria:

* Inability to provide informed consent
* Pregnant, breastfeeding, or planning for either in the next 6 months or <6 months postpartum
* Low C-peptide and possible subsequent GAD 65 level that suggests type 1 diabetes, clinical factors that suggest type 1 diabetes (lean, lack of family history, and diabetic ketoacidosis in the past) or a previous diagnosis of type 1 diabetes or latent autoimmune diabetes
* Cancer, heart failure, or kidney failure
* Vegan
* Untreated mental health condition
* Currently following a very low-carbohydrate diet or breakfasts
* Thyroid levels out of range
* Alcoholism
* Previous bariatric surgery
* Difficulty chewing or swallowing
* Dependence on others for food preparation
* Currently enrolled in another investigative study that might conflict with this research

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-10-17 (Actual)

PRIMARY OUTCOMES:
Intervention satisfaction | At 4 months
  A 1-item measure about intervention satisfaction. We ask participants, "How would you rate your overall satisfaction with the program?" The item is rated from 1 = very dissatisfied to 6 = very satisfied, with higher scores reflecting greater satisfaction.

SECONDARY OUTCOMES:
Weekly dietary adherence | Weekly over 4 months
  A 1-item measure about dietary adherence. We ask participants to reflect on the past week and rate whether they ate a low-carbohydrate breakfast. The item is rated from 1 = not at all to 7 = very much so, with higher scores reflecting greater adherence.
Change in diabetes treatment satisfaction | 0 to 4 months
  The Diabetes Treatment Satisfaction Questionnaire is an 8-item measure of satisfaction with current diabetes therapy over the past several weeks. Each item is rated on a 7-point scale. Six items form the Treatment Satisfaction scale, assessing overall satisfaction, perceived convenience and flexibility, understanding of diabetes, and willingness to recommend or continue the current regimen. Two additional items evaluate the perceived frequency of unacceptable hyperglycemia and hypoglycemia. The Treatment Satisfaction score is calculated from the six satisfaction items, with higher scores indicating greater satisfaction; the two frequency items are scored separately, with higher values reflecting more frequent high or low blood glucose levels.
Change in health-related quality of life | 0 to 4 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS)-29 is a 29-item survey for assessing health-related quality of life across seven domains (Physical function, Anxiety, Depression, Fatigue, Sleep disturbance, Social roles, and Pain interference) plus Pain intensity. All domains are scored using T-scores (mean 50, SD 10), where higher scores indicate better function for functional domains (Physical Function, Social Roles) and worse symptoms for symptom domains (Anxiety, Depression, Fatigue, Sleep Disturbance, Pain Interference).
Change in HbA1c | 0 to 4 months
  This will assess the change in the level reported for this outcome
Change in anti-hyperglycemic medications | 0 to 4 months
  The Medication Effect Score (MES) quantifies the overall intensity of antiglycemic therapy, with higher scores indicating greater medication requirements. For each diabetes medication, the percentage of the maximum recommended daily dose is multiplied by an adjustment factor reflecting its expected hemoglobin A1c-lowering potency; these values are summed to yield the total MES. Scores range from 0 upward (no fixed maximum), with lower scores reflecting lower medication intensity.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hansen A, Raymond K, Simon A, Kim S, Bayandorian H, Marriott D, Saslow LR. Very Low-Carbohydrate Breakfast Intervention for Adults with Type 2 Diabetes and Persistent Hyperglycemia: Protocol for a Digital, Nonrandomized Pre-Post Study. JMIR Res Protoc. 2026 Jan 28;15:e81041. doi: 10.2196/81041. PMID 41605502

DOCUMENTS (1):
  • Informed Consent Form (2024-11-14): https://cdn.clinicaltrials.gov/large-docs/97/NCT05986097/ICF_000.pdf